CLINICAL TRIAL: NCT04767854
Title: Digital Osteoarthritis Care- DigiOA
Brief Title: Digital Osteoarthritis Care
Acronym: DigiOA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: The Dam Foundation (Other); The Norwegian Council for Musculoskeletal Health (Unknown)
Responsible Party: Principal Investigator, Anne Therese Tveter, Principal Investigator, Assosiate Professor, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/FO347383
Record Dates: First submitted 2021-02-15; First posted 2021-02-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Telerehabilitation; Digital care; mHealth
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OA school + Virtual Training mobile health application (Experimental): After a clinical examination by the physiotherapist, all patients will receive a 1-2-hour group session of patient education according to guidelines.
  The intervention group will receive an individually tailored exercise program through the Virtual Training mobile health application. After each exercise the patient score his/her execution of the exercise on a Likert-scale of 1 to 5, judging their effort from very poor to very good. After the session, patients rate their pain on a Numeric Rating Scale from 0 to 10. The patients in the intervention group will be instructed to exercise 3 times per week for 6 weeks. If the patients want to exercise more than 3 times per week, the exercise program will be available in the app once every day.
  Interventions: Behavioral: OA school; Other: Virtual Training mobile health application
- OA school + usual care (Active Comparator): After a clinical examination by the physiotherapist, all patients will receive a 1-2-hour group session of patient education according to guidelines.
  The control group will receive individually tailored supervised exercise therapy by a physiotherapist individually or in a group setting, twice a week for 6 weeks. Additionally, the patients will be motivated to perform one session of home exercise a week, a total of 3 sessions per week
  Interventions: Behavioral: OA school; Other: Usual care

INTERVENTIONS:
Behavioral: OA school — Patient education according to guidelines, with information about e.g. disease progression, symptoms, treatment, exercise, self-care techniques and dietary information
Other: Virtual Training mobile health application — Individually tailored home exercise programs delivered through a mobile health application
  Arms: OA school + Virtual Training mobile health application
Other: Usual care — Individually tailored exercise programs conducted in weekly supervised individual or group sessions
  Arms: OA school + usual care

SUMMARY:
Osteoarthritis (OA) is among the most prevalent and costly diseases, with an estimate of $460 billion in all-cause medical costs. It causes pain and reduced physical function, and with no existing cure, the recommended first-line treatment is information, exercise and weight management if indicated. As the prevalence of OA is expected to increase in the coming years, exploring innovative solutions to maintain economical sustainable treatment in the future becomes a necessity. Telerehabilitation, technology which involves providing treatment through information and communication technology, regardless of the patient's geographical location, has shown its potential within cardiac, pulmonary, neurological and musculoskeletal conditions.

Virtual Training (VT) is a generic mobile health application used to deliver digital home exercise programs with text, audio and video support. Through a novel feedback system the therapist is able monitor the patients progress and pain level during exercise. This project aims to investigate, through a randomized controlled trial (RCT), whether the use of the VT-app is as effective as supervised exercise therapy in improving pain, physical function and disease activity in patients with hip and/or knee osteoarthritis. In addition, the investigators want to investigate if the use of the app is more cost effective than supervised exercise therapy, whether the use increases adherence with first line treatment, and whether there are certain characteristics of the patients responding to the intervention.

DETAILED DESCRIPTION:
The study is a two-armed non-inferiority randomized controlled trial (RCT) situated in the primary care setting in Norway. Participants diagnosed with hip and/or knee OA will be randomized to either exercise therapy via app or usual care. Patients aged 18 years and older presenting with activity-related hip and/or knee pain/complaints and clinical signs and symptoms corresponding to hip and/or knee OA seeking treatment at physiotherapist working in private practice, will be included if eligible for the study.

The research questions are:

1. Is exercise therapy, delivered through a mobile health application (Virtual Training), as effective as supervised exercise therapy in patients with hip and/or knee OA, measured by number of patients classified as responders according to the OMERACT-OARSI responder criteria?
2. Is exercise therapy delivered through Virtual Training more cost-effective regarding health care and medication use than supervised exercise therapy for patients with hip and/or knee OA?
3. Will patients with hip and/or knee OA, using Virtual Training, be more adherent to exercise during the intervention period compared to patients undergoing supervised exercise therapy, and are there any demographic or clinical factors characterizing the OMERACT-OARSI responding patients using Virtual Training?

The primary analysis will be conducted on an intention-to-treat basis by comparing the proportion of responders at 6 weeks and 3 months post-intervention according to the OMERACT-OARSI responder criteria in the intervention and the control group using logistic regression analysis. Per-protocol analyses will also be conducted. Difference in secondary outcomes will be assessed using analysis of covariance (ANCOVA) on the post-intervention values, with baseline values as covariates.

Cost-effectiveness will be evaluated assessing the difference in health care and medication use and quality of life during 3-month follow-up, reporting the incremental cost-effectiveness ratio (ICER) reflecting the between-group difference in incremental cost per adjusted life years (QALYs). Between-group difference in adherence to exercise will be assessed using linear regression, while patient characteristics in the intervention group will be assessed using logistic regression. Additional analyses assessing associations between physical activity, efficacy, barriers for exercise and OA-related questions will also be assessed in secondary analyses.

ELIGIBILITY:
Inclusion Criteria:

* Activity-related hip and/or knee pain/complaints and clinical signs and symptoms corresponding to hip and/or knee OA
* Access to smartphone or tablet

Exclusion Criteria:

* Neurological disorders
* Contraindication to physical activity
* Total hip or knee replacement in the actual joint(s) with no pain/ complaints in the other hip or knee joint(s)
* Inflammatory rheumatic diseases (e.g. rheumatoid arthritis, spondyloarthritis)
* Malignant illness or other major conditions (e.g. unstable cardiovascular disorders or lung disease, dementia) that restrict the ability to adhere to the recommended treatment
* Not understanding the Norwegian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of responders according to OMERACT-OARSI responder criteria | 6 weeks (end of intervention period)
  A patient is classified as a responder if one of the following criteria is fulfilled:
  1. High improvement in pain or function from baseline to follow-up
     * ≥50% improvement + absolute change of ≥2 in pain, OR
     * ≥50% improvement + absolute change of ≥2 in function
  2. Improvement in at least two of the three following from baseline to follow-up:
     * ≥20% improvement + absolute change ≥1 in pain
     * ≥20% improvement + absolute change ≥1 in function
     * ≥20% improvement + absolute change ≥1 in the patient´s global assessment of disease activity

SECONDARY OUTCOMES:
Number of responders according to OMERACT-OARSI responder criteria | 18 weeks post randomization
  A patient is classified as a responder if one of the following criteria is fulfilled:
  1. High improvement in pain or function from baseline to follow-up
     * ≥50% improvement + absolute change of ≥2 in pain, OR
     * ≥50% improvement + absolute change of ≥2 in function
  2. Improvement in at least two of the three following from baseline to follow-up:
     * ≥20% improvement + absolute change ≥1 in pain
     * ≥20% improvement + absolute change ≥1 in function
     * ≥20% improvement + absolute change ≥1 in the patient´s global assessment of disease activity
Physical performance test, 30 seconds sit to stand test (30 sec STS) | Baseline
  Number of repetitions in the 30 seconds sit to stand-test
Physical performance test, 30 seconds sit to stand test (30 sec STS) | 6 weeks (end of intervention period)
  Number of repetitions in the 30 seconds sit to stand-test
Self reported goal achievement, Patient-specific functional scale (PSFS) | Baseline
  Patients will address one to three activities they have problems performing due to osteoarthritis. The degree of difficulty with performing these activities is rated from 0 (cannot perform the activity) to 10 (no problems)
Self reported goal achievement, Patient-specific functional scale (PSFS) | 6 weeks (end of intervention period)
  Patients will address one to three activities they have problems performing due to osteoarthritis. The degree of difficulty with performing these activities is rated from 0 (cannot perform the activity) to 10 (no problems)
Self reported goal achievement, Patient-specific functional scale (PSFS) | 18 weeks post randomization
  Patients will address one to three activities they have problems performing due to osteoarthritis. The degree of difficulty with performing these activities is rated from 0 (cannot perform the activity) to 10 (no problems)
Hip pain and function, Hip disability and Osteoarthritis Outcome Score (HOOS) | Baseline
  Result in the last week disability on five subscales; pain (10 items, scale 0-40), symptoms (5 items, scale 0-20), function in daily living (17 items, scale 0-68), function in sport and recreation (4 items, scale 0-16) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability)
Hip pain and function, Hip disability and Osteoarthritis Outcome Score (HOOS) | 6 weeks (end of intervention period)
  Result in the last week disability on five subscales; pain (10 items, scale 0-40), symptoms (5 items, scale 0-20), function in daily living (17 items, scale 0-68), function in sport and recreation (4 items, scale 0-16) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability)
Hip pain and function, Hip disability and Osteoarthritis Outcome Score (HOOS) | 18 weeks post randomization
  Result in the last week disability on five subscales; pain (10 items, scale 0-40), symptoms (5 items, scale 0-20), function in daily living (17 items, scale 0-68), function in sport and recreation (4 items, scale 0-16) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability)
Knee pain and function, Knee disability and Osteoarthritis Outcome Score (KOOS) | Baseline
  Result in the last week disability on five subscales; pain (9 items, scale 0-36), symptoms (7 items, scale 0-28), function in daily living (17 items, scale 0-68), function in sport and recreation (5 items, scale 0-20) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability)
Knee pain and function, Knee disability and Osteoarthritis Outcome Score (KOOS) | 6 weeks (end of intervention period)
  Result in the last week disability on five subscales; pain (9 items, scale 0-36), symptoms (7 items, scale 0-28), function in daily living (17 items, scale 0-68), function in sport and recreation (5 items, scale 0-20) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability)
Knee pain and function, Knee disability and Osteoarthritis Outcome Score (KOOS) | 18 weeks post randomization
  Result in the last week disability on five subscales; pain (9 items, scale 0-36), symptoms (7 items, scale 0-28), function in daily living (17 items, scale 0-68), function in sport and recreation (5 items, scale 0-20) and quality of life (4 items, scale 0-16). Items are scored by a five-point Likert scale ranging from 0 (least severe) to 4 (most severe). Total sum-score and subscale sum-scores will be converted to normalized scores ranging from 0 (extreme disability) to 100 (no disability)
Self-reported physical activity, International Physical Activity Questionnaire-Short Form (IPAQ) | Baseline
  Measured by The International Physical Activity Questionnaire-Short Form: Amount of time (minutes per week/day) spent on sitting, walking, and moderate- and vigorous intensity physical activity the last week (0-7 days). Results are reported as MET-scores and are categorized into categorical score of low, moderate or high level of physical activity.
Self-reported physical activity, International Physical Activity Questionnaire-Short Form (IPAQ) | 6 weeks (end of intervention)
  Measured by The International Physical Activity Questionnaire-Short Form: Amount of time (minutes per week/day) spent on sitting, walking, and moderate- and vigorous intensity physical activity the last week (0-7 days). Results are reported as MET-scores and are categorized into categorical score of low, moderate or high level of physical activity.
Self-reported physical activity, International Physical Activity Questionnaire-Short Form (IPAQ) | 18 weeks post randomization
  Measured by The International Physical Activity Questionnaire-Short Form: Amount of time (minutes per week/day) spent on sitting, walking, and moderate- and vigorous intensity physical activity the last week (0-7 days). Results are reported as MET-scores and are categorized into categorical score of low, moderate or high level of physical activity.
Self-reported self-efficacy, Arthritis Self-Efficacy Scale (ASES) | Baseline
  Measured by Arthritis Self-Efficacy Scale: average score in the subelements pain (5 questions) and symptoms (6 questions) on a 5 point Likert scale (very uncertain to very sure). Higher average score indicate higher degree of self-efficacy.
Self-reported self-efficacy, Arthritis Self-Efficacy Scale (ASES) | 6 weeks (end of intervention)
  Measured by Arthritis Self-Efficacy Scale: average score in the subelements pain (5 questions) and symptoms (6 questions) on a 5 point Likert scale (very uncertain to very sure). Higher average score indicate higher degree of self-efficacy.
Self-reported self-efficacy, Arthritis Self-Efficacy Scale (ASES) | 18 weeks post randomization
  Measured by Arthritis Self-Efficacy Scale: average score in the subelements pain (5 questions) and symptoms (6 questions) on a 5 point Likert scale (very uncertain to very sure). Higher average score indicate higher degree of self-efficacy.
Exercise self-efficacy | Baseline
  Measured by the Exercise self-efficacy scale containing the subscales self-efficacy for exercise, barriers to exercise, benefits of exercise and the impact of exercise on OA. Each subscale contains 3-8 questions relevant to the topic, with a 5-point Likert scale ranging from strongly disagree to strongly agree. A sum score of the subscales is calculated, ranging from 20 to 100, with higher scores indicating less barriers and greater self-efficacy with physical activity.
Exercise self-efficacy | 6 weeks (end of intervention)
  Measured by the Exercise self-efficacy scale containing the subscales self-efficacy for exercise, barriers to exercise, benefits of exercise and the impact of exercise on OA. Each subscale contains 3-8 questions relevant to the topic, with a 5-point Likert scale ranging from strongly disagree to strongly agree. A sum score of the subscales is calculated, ranging from 20 to 100, with higher scores indicating less barriers and greater self-efficacy with physical activity.
Exercise self-efficacy | 18 weeks post randomization
  Measured by the Exercise self-efficacy scale containing the subscales self-efficacy for exercise, barriers to exercise, benefits of exercise and the impact of exercise on OA. Each subscale contains 3-8 questions relevant to the topic, with a 5-point Likert scale ranging from strongly disagree to strongly agree. A sum score of the subscales is calculated, ranging from 20 to 100, with higher scores indicating less barriers and greater self-efficacy with physical activity.
Health-related quality of life, EuroQoL (EQ5D-5L) | Baseline
  Health-related quality of life is measured by the EQ5D-5L questionnaire. Patients are asked to answer their ability to perform walking, personal care and activities of daily life on a 5 point Likert scale from no difficulties to not able to. Pain and anxiety/depression is measured on a 5 point Likert scale from no pain to very strong pain, and no anxiety/depression to extremely anxious/depressed. General experience of health is measured from 0 (worst health) to 100 (best health) on a numeric rating scale.
Health-related quality of life, EuroQoL (EQ5D-5L) | 6 weeks (end of intervention)
  Health-related quality of life is measured by the EQ5D-5L questionnaire. Patients are asked to answer their ability to perform walking, personal care and activities of daily life on a 5 point Likert scale from no difficulties to not able to. Pain and anxiety/depression is measured on a 5 point Likert scale from no pain to very strong pain, and no anxiety/depression to extremely anxious/depressed. General experience of health is measured from 0 (worst health) to 100 (best health) on a numeric rating scale.
Health-related quality of life, EuroQoL (EQ5D-5L) | 18 weeks post randomization
  Health-related quality of life is measured by the EQ5D-5L questionnaire. Patients are asked to answer their ability to perform walking, personal care and activities of daily life on a 5 point Likert scale from no difficulties to not able to. Pain and anxiety/depression is measured on a 5 point Likert scale from no pain to very strong pain, and no anxiety/depression to extremely anxious/depressed. General experience of health is measured from 0 (worst health) to 100 (best health) on a numeric rating scale.
Anxiety and depression, Hopkins symptom checklist (HSCL-5) | Baseline
  Symptoms of anxiety and depression is measured by the short form of the Hopkins symptom checklist. Patients answers on five statements is used to measure general symptoms of anxiety and depression from the last 14 days, answers ranging from Not at all to Very much. Total sum score is (0-20) is calculated, higher score indicating greater symptoms of anxiety and depression.
Anxiety and depression, Hopkins symptom checklist (HSCL-5) | 6 weeks (end of intervention)
  Symptoms of anxiety and depression is measured by the short form of the Hopkins symptom checklist. Patients answers on five statements is used to measure general symptoms of anxiety and depression from the last 14 days, answers ranging from Not at all to Very much. Total sum score is (0-20) is calculated, higher score indicating greater symptoms of anxiety and depression.
Anxiety and depression, Hopkins symptom checklist (HSCL-5) | 18 weeks post randomization
  Symptoms of anxiety and depression is measured by the short form of the Hopkins symptom checklist. Patients answers on five statements is used to measure general symptoms of anxiety and depression from the last 14 days, answers ranging from Not at all to Very much. Total sum score is (0-20) is calculated, higher score indicating greater symptoms of anxiety and depression.
Social participation | Baseline
  Limitations in social activities or contact with family, friends, neighbours or others last 14 days is reported on the social participation-subscale of the COOP/WONCA Functional Assessments Charts. Reported on a 5 point Likert scale ranging from Not at all to Very much, with Very much indicating greater limitations in social contact.
Social participation | 6 weeks (end of intervention)
  Limitations in social activities or contact with family, friends, neighbours or others last 14 days is reported on the social participation-subscale of the COOP/WONCA Functional Assessments Charts. Reported on a 5 point Likert scale ranging from Not at all to Very much, with Very much indicating greater limitations in social contact.
Social participation | 18 weeks post randomization
  Limitations in social activities or contact with family, friends, neighbours or others last 14 days is reported on the social participation-subscale of the COOP/WONCA Functional Assessments Charts. Reported on a 5 point Likert scale ranging from Not at all to Very much, with Very much indicating greater limitations in social contact.
Usability of mobile health application, System Usability Scale (SUS) | 6 weeks (end of intervention)
  Usability of the Virtual Training health application for patients, measured by the System Usability Scale. 10 item questionnaire with five response options for respondents; from strongly agree to strongly disagree
Usage of medication | Baseline
  Usage of medications last three months. Measured in dosage and frequency.
Usage of medication | 18 weeks post randomization
  Usage of medications last three months. Measured in dosage and frequency.
Change in disease activity | Baseline and 6 weeks (end of intervention)
  Change in disease activity from baseline is reported on a 7 point Likert scale rating from Very much worse to Very much better.
Change in disease activity | Baseline and 18 weeks post randomization
  Change in disease activity from baseline is reported on a 7 point Likert scale rating from Very much worse to Very much better.
Disease activity | Baseline
  Last week's experience of disease activity is measured on a Numeric rating scale ranging from 0 (Good, no symptoms) to 10 (Very bad).
Disease activity | 6 weeks (end of intervention)
  Last week's experience of disease activity is measured on a Numeric rating scale ranging from 0 (Good, no symptoms) to 10 (Very bad).
Disease activity | 18 weeks post randomization
  Last week's experience of disease activity is measured on a Numeric rating scale ranging from 0 (Good, no symptoms) to 10 (Very bad).
Diagnose specific pain experience | Baseline
  Last week's experience of pain is measured on a Numeric rating scale ranging from 0 (No pain) to 10 (Worst imaginable pain).
Diagnose specific pain experience | 6 weeks (end of intervention)
  Last week's experience of pain is measured on a Numeric rating scale ranging from 0 (No pain) to 10 (Worst imaginable pain).
Diagnose specific pain experience | 18 weeks post randomization
  Last week's experience of pain is measured on a Numeric rating scale ranging from 0 (No pain) to 10 (Worst imaginable pain).
Fatigue | Baseline
  Last week's experience of fatigue is measured on a Numeric rating scale from 0 (No fatigue) to 10 (Worst imaginable fatigue).
Fatigue | 6 weeks (end of intervention)
  Last week's experience of fatigue is measured on a Numeric rating scale from 0 (No fatigue) to 10 (Worst imaginable fatigue).
Fatigue | 18 weeks post randomization
  Last week's experience of fatigue is measured on a Numeric rating scale from 0 (No fatigue) to 10 (Worst imaginable fatigue).
Use of health care services | 6 weeks (end of intervention)
  Usage of health care services is measured by number of consultations to general practioner, medical specialist, physical therapist, occupational therapist and Healthy Life Centres, and number of x-rays and MRI's undertaken, last six weeks.
Use of health care services | 18 weeks post randomization
  Usage of health care services is measured by number of consultations to general practioner, medical specialist, physical therapist, occupational therapist and Healthy Life Centres, and number of x-rays and MRI's undertaken, last three months.
General digital competence | Baseline
  19 questions concerning general digital competence, evaluated on a 4 point Likert-scale ranging from very difficult to very easy. Included also an option of answering Don't know.
Satisfaction with use of app in exercise therapy | 6 weeks (end of intervention)
  Satisfaction with use of app in exercise therapy evaluated on a visual analog scale ranging from very little satisfied to very satisfied (0-10). Question only concerns patients in intervention arm.
Suitability of using an app in exercise therapy | 6 weeks (end of intervention)
  Suitability of using an app in exercise therapy evaluated on a visual analog scale ranging from very unsuitable to very suitable (0-10). Question only concerns patients in intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Therese Tveter, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (13):
- Norway (13):
  - Laguneparken fysioterapi/Arna fysikalske, Bergen
  - Sandviken fysioterapi og trening, Bergen
  - Trimmen, Drammen
  - Sentrum Fysioterapi, Gjøvik
  - Ace Treningssenter, Indre Østfold
  - Trøgstad fysioterapi, Indre Østfold
  - Nittedal fysikalske institutt, Nittedal
  - Physiotherapist Stein Listaul, Notodden
  - Aktifys Institutt, Oslo
  - Furuset Fysioterapi, Oslo
  - Røa Centrum Fysioterapi og Akupunktur, Oslo
  - Ski Fysioterapisenter, Ski
  - Skiptvet Fysikalske, Skiptvet

IPD SHARING:
Plan to Share IPD: No
Data may be made available on reasonably request to principal investigator

REFERENCES:
- [Derived] Martinsen L, Osteras N, Moseng T, Tveter AT. Adherence to in-person and app-based exercise for patients with hip or knee osteoarthritis; secondary analyses from a randomized controlled trial. Rheumatol Int. 2025 Aug 26;45(9):208. doi: 10.1007/s00296-025-05967-4. PMID 40856813
- [Derived] Martinsen L, Osteras N, Moseng T, Tveter AT. Effect of a mHealth exercise intervention compared with supervised exercise therapy in osteoarthritis management: protocol of the DigiOA trial. BMJ Open. 2022 Sep 23;12(9):e066248. doi: 10.1136/bmjopen-2022-066248. PMID 36153027

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT04767854/SAP_000.pdf